CLINICAL TRIAL: NCT01580514
Title: Cardioprotective Effects of Exenatide in Patients With ST-segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention ; Results of Exenatide Myocardial Protection In REvascularization (EMPIRE) Study
Brief Title: Myocardial Protection of Exenatide in AMI
Acronym: EMPIRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Weon Kim, associate professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHMC-2012001
Record Dates: First submitted 2012-04-13; First posted 2012-04-19 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; percutaneous coronary intervention; exenatide; reperfusion injury; cardiac magnetic resonance
MeSH Terms: conditions — Myocardial Infarction; Reperfusion Injury | interventions — Sodium Chloride; Exenatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide (Active Comparator): Drug: Exenatide
  10 μg subcutaneous and 10 μg intravenously injection of exenatide BYETTA® (Amylin-Lilly) 5 min before the onset of reperfusion. And twice daily 10 μg subcutaneous injection was continued on the following 2 days.
  Interventions: Drug: exenatide BYETTA® (Amylin-Lilly)
- Saline (Placebo Comparator): Drug: Saline
  10 μg subcutaneous and 10 μg intravenously injection of equivalent volume of normal saline 5 min before the onset of reperfusion. And twice daily 10 μg subcutaneous injection was continued on the following 2 days.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: exenatide BYETTA® (Amylin-Lilly) — After informed consent was obtained, patients who met the enrollment criteria were randomly assigned to either the control group or the exenatide group.
  Patients assigned to exenatide were treated with 10 μg subcutaneous and 10 μg intravenously injection of exenatide BYETTA® (Amylin-Lilly) 5 min before the onset of reperfusion. And twice daily 10 μg subcutaneous injection was continued on the following 2 days.
  Other Names: Saline
  Arms: Exenatide
Drug: Saline — After informed consent was obtained, patients who met the enrollment criteria were randomly assigned to either the control group or the exenatide group.
  Patients assigned to saline were treated with 10 μg subcutaneous and 10 μg intravenously injection of equivalent volume of normal saline 5 min before the onset of reperfusion. And twice daily 10 μg subcutaneous injection was continued on the following 2 days.
  Other Names: Exenatide
  Arms: Saline

SUMMARY:
Experimental evidence suggests exenatide, a glucagon-like peptide 1 receptor analogue, has significant cardiovascular protective effects in various conditions. The investigators examined whether conventional use of exenatide at the time of primary percutaneous coronary intervention would reduce the infarct size in patients with ST-segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
In this proof-of-concept trial, we assessed the effects of acute-phase adjunctive exenatide therapy in patients with STEMI.

Infarct size after STEMI was evaluated by both cardiac magnetic resonance image and cardiac biomarkers compared with standard treatment.

LV function was assessed by conventional and speckle tracking echocardiography. During 6-month follow up, the safety/tolerability of exenatide and clinical outcomes were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 79 years
* patients presenting with first ST-segment elevation myocardial infarction
* Thrombolysis in Myocardial Infarction [TIMI] flow grade 0)

Exclusion Criteria:

* cardiac arrest
* ventricular fibrillation
* cardiogenic shock
* hemodynamic instability
* suspicious stent thrombosis
* left bundle branch block
* previous acute myocardial infarction
* previous coronary artery bypass operation
* significant valvular heart disease
* primary myocardial disease
* atrial fibrillation
* significant hepatic or renal dysfunction, hypoglycaemia,
* diabetic ketoacidosis
* active infection or chronic inflammatory disease
* malignancy
* women who were pregnant or who were of childbearing age

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Infarct size | 1 month
  Infarct size was assessed by measuring the release of creatine kinase-MB and troponin I during 72 hours and by performing cardiac magnetic resonance imaging on 1 month after infarction.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 6 month after primary PCI
  Adverse events of exenatide such as hypoglycemia, nausea, vomiting, and chest pain aggravation were monitored during study period.
LV function | at admission and 6 month after primary PCI
  Conventional and speckle tracking echocardiography was performed at initial presentation and 3 days and 6 months after primary PCI.
Clinical outcomes | 6 months after primary PCI
  During 6-month follow up, clinical outcomes such as all death, repeated myocardial infarction or repeated PCI were also assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Weon Kim, MD, PhD, Principal Investigator — Division of Cardiology, Department of Internal Medicine, Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Timmers L, Henriques JP, de Kleijn DP, Devries JH, Kemperman H, Steendijk P, Verlaan CW, Kerver M, Piek JJ, Doevendans PA, Pasterkamp G, Hoefer IE. Exenatide reduces infarct size and improves cardiac function in a porcine model of ischemia and reperfusion injury. J Am Coll Cardiol. 2009 Feb 10;53(6):501-10. doi: 10.1016/j.jacc.2008.10.033. PMID 19195607
- [Derived] Huang M, Wei R, Wang Y, Su T, Li Q, Yang X, Chen X. Protective effect of glucagon-like peptide-1 agents on reperfusion injury for acute myocardial infarction: a meta-analysis of randomized controlled trials. Ann Med. 2017 Nov;49(7):552-561. doi: 10.1080/07853890.2017.1306653. Epub 2017 Mar 31. PMID 28286967
- [Derived] Woo JS, Kim W, Ha SJ, Kim JB, Kim SJ, Kim WS, Seon HJ, Kim KS. Cardioprotective effects of exenatide in patients with ST-segment-elevation myocardial infarction undergoing primary percutaneous coronary intervention: results of exenatide myocardial protection in revascularization study. Arterioscler Thromb Vasc Biol. 2013 Sep;33(9):2252-60. doi: 10.1161/ATVBAHA.113.301586. Epub 2013 Jul 18. PMID 23868944